CLINICAL TRIAL: NCT01739400
Title: Long Term, Single-arm, Open-label Extension Study of Protocol AC-055-305 to Assess the Safety, Tolerability and Efficacy of Macitentan in Subjects With Eisenmenger Syndrome
Brief Title: Clinical Study to Assess the Long-term Safety, Tolerability, and Efficacy of Macitentan in Subjects With Eisenmenger Syndrome
Acronym: MAESTRO-OL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary endpoint of parent study AC-055-305/MAESTRO (NCT01743001) not met.
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-308
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Eisenmenger Syndrome; exercise capacity
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Eisenmenger Complex | interventions — macitentan; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Macitentan (Experimental): Macitentan 10 mg tablet, once daily.
  Interventions: Drug: Macitentan 10 mg tablet, once daily.

INTERVENTIONS:
Drug: Macitentan 10 mg tablet, once daily. — Macitentan 10 mg tablet, once daily.
  Other Names: Macitentan; ACT-064992

SUMMARY:
Long-term study to evaluate if macitentan is safe, tolerable and efficient enough to be used for treatment of Eisenmenger syndrome.

ELIGIBILITY:
Inclusion Criteria:

Subjects with ES (including those with Down Syndrome) having completed the double-blind AC-055-305 / MAESTRO study as scheduled, i.e., who remained in the double-blind study up to Week 16 (whether or not they were still taking study drug at the end of this period).

Exclusion Criteria:

Subjects who prematurely discontinue double-blind study drug during the AC-055-305 / MAESTRO study due to:

* an AE assessed as related to the use of study drug,
* or elevated liver tests (related or unrelated to study drug).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (5):
  - Emory University Hospital/the Emory Clinic, Atlanta, Georgia
  - Barnes-Jewish Hosp/Wash Univ School of Med, St Louis, Missouri
  - Children'S Heart Center Nevada, Las Vegas, Nevada
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Children'S Hosp - Dept of Cardiology, Houston, Texas
- Gen Hosp Univ Vienna Dept Cardiology, Vienna, Austria
- Bulgaria (3):
  - Mhat Nat Card Hosp - Cardiology Clinic, Sofia
  - Mhat Nat Card Hosp - Pediatric Clin / Ped Card Dept, Sofia
  - Mhat Sveta Anna Clin Card, Sofia
- Chile (2):
  - Instituto Nacional del Torax, Providencia, Santiago RCH
  - Clinica Tabancura - Cardio Unit, Santiago
- China (6):
  - Guangdong General Hospital, Cardiology Dpt, Guangzhou, Guangdong
  - Wu Han Asia Heart Hosp, Wuhan, Hubei
  - The General Hosp of Shenyang Military Region, Shenyang, Liaoning
  - Beijing Anzhen Hospital, Cardiology Dpt, Beijing
  - Cardiovascular Institute&Fuwai Hospital, Beijing
  - Shanghai Pulmonary Hospital, Dept of Pulmonary Circulation, Shanghai
- France (4):
  - Hosp La Timone - Dept Pediatric Cardiology, Marseille
  - Hosp Laennec - Dept Cardiology, Nantes
  - Hosp Pompidou - Dept Congenital Cardiac Diseases, Paris
  - Hosp Cardiology Haut Leveque - Dept Congenital Diseases, Pessac
- Germany (3):
  - Herzzentrum Berlin, Ped Cardiology, Berlin
  - Universitätsklinikum Giessen - Pediatric Heart Center, Giessen
  - Uni Heidelberg - Kinderkardiologie, Heidelberg
- Ahepa University General Hospital, Thessaloniki, Greece
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Mexico (3):
  - Unidad de Investigacion Clin En Med, Sc (Udicem), Monterrey, Nuevo León
  - Instituto Nacional de Cardiologia (Inc) Ignacio Chavez, Mexico City
  - Instituto de Corazon de Querètaro, Querétaro
- PHC, MAB, Manila, Philippines
- Poland (3):
  - Cardiology Gdańsk Univ, Gdansk
  - Cardiology Kraków Univ, Krakow
  - Cardiology Wrocław, Wroclaw
- Portugal (2):
  - Hosp Univ Coimbra - Dpt Cardiology, Coimbra
  - Hosp Sta Marta - Dept Cardiology, Lisbon
- Romania (3):
  - Er Inst For Cardvasc Dis "Prof Dr Cc Iliescu" - Card Ii, Bucaresti
  - Cardio Med Srl, Târgu Mureş
  - Clin Hosp For Inf and Pulm Dis Victor Babes - Ii Pulm, Timișoara
- Russia (3):
  - Sci Institute Systemic Poriblems Cardio Diseases Kemerovo, Kemerovo
  - Russian Cardiology Scientific and Production Complex, Moscow
  - V. A. Almazov Institute of Cardiology, Saint Petersburg
- Serbia (3):
  - Dedinje Cardiovasc Inst - Cardiovasc Research Ctr, Belgrade
  - Mother and Child Health Care Institute Dr. Vukan Cupic, Belgrade
  - Clin Hosp Ctr Zemun - Cardiology Dept, Belgrade
- Spain (3):
  - Hosp Univ Vall D'Hebron - Dpt Congenital Heart Disease Adult, Barcelona
  - Hosp Univ Virgen Macarena - Dpt Cardiology, Seville
  - Hosp Universitario La Fe Dpt Cardiology, Valencia
- Bristol Univ Hosp Congenital Heart Centre, Bristol, United Kingdom
- Vietnam (3):
  - Hanoi Medical University Hospital, Hanoi
  - Children'S Hospital, Ho Chi Minh, Ho Chi Minh City
  - Tam Duc Hospital, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 51 sites in 19 countries (geographical regions: Asia-Pacific, Eastern Europe, Latin America, North America and Western Europe).
Pre-assignment Details: 217 of 221 subjects (111 macitentan, 110 placebo) that completed treatment in the AC-055-305/MAESTRO double-blind (DB) parent study (NCT01743001) were enrolled in the open-label (OL) study without knowledge of their study treatment allocation in the DB study (macitentan or placebo).
Groups:
- DB-macitentan: All subjects treated with macitentan in the DB study (AC-055-305, NCT01743001).
- DB-placebo: All subjects treated with placebo in the DB study (AC-055-305, NCT01743001).
Period: Overall Study
Arm/Group | DB-macitentan | DB-placebo
Started (Enrolled from DB parent study MAESTRO (AC-0553-305, NCT01743001)) | 109 | 108
Treated With 10 mg Macitentan | 109 | 108
Completed (Completed OL study) | 92 | 99
Not Completed | 17 | 9
Not completed — Physician Decision | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 5 | 2
Not completed — Withdrawal by Subject | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- DB-macitentan: All enrolled subjects treated with macitentan in the AC-055-308 / OL study who received macitentan in the DB study (AC-055-305, NCT01743001).
- DB-placebo: All enrolled subjects treated with macitentan in the AC-055-308 / OL study who received placebo in the DB study (AC-055-305, NCT01743001).
- Total: Total of all reporting groups
Arm/Group | DB-macitentan | DB-placebo | Total
Number analyzed (Participants) | 109 | 108 | 217
Age, Continuous [Mean (Full Range); unit: years] | 34.6 [12 to 82] | 34.6 [14 to 62] | 34.6 [12 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 66 | 143
  Male | 32 | 42 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89 | 88 | 177
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 52 | 51 | 103
  Chinese | 35 | 35 | 70
  Other Asian | 11 | 11 | 22
  Other | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Asia-Pacific: Asia-Pacific | 45 | 44 | 89
  Asia-Pacific: Eastern Europe | 24 | 26 | 50
  Asia-Pacific: Latin America | 18 | 18 | 36
  Asia-Pacific: North America | 1 | 4 | 5
  Asia-Pacific: Western Europe-Israel | 21 | 16 | 37
Age categorical [Count of Participants; unit: Participants]
  12 - 17 years | 12 | 2 | 14
  18 - 55 years | 89 | 99 | 188
  ≥ 56 years | 8 | 7 | 15
WHO Functional Class (FC) [Count of Participants; unit: Participants] — WHO functional class of subjects Class I: no symptoms with exercise or at rest. No limitation of activity. Class II: No symptoms at rest but slight limitation with ordinary activities causing symptoms (e.g. short of breath with climbing a flight of stairs, grocery shopping, or making the bed). Class III: may not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. Class IV: symptoms at rest (e.g. dyspnea and/or fatigue) and inability to carry out any physical activity without symptoms. Patients in class IV manifest signs of right heart failure
  Participants
    Class I | 0 | 0 | 0
    Class II | 66 | 65 | 131
    Class III | 43 | 43 | 86
    Class IV | 0 | 0 | 0
Downs syndrome status [Count of Participants; unit: Participants]
  Yes | 10 | 10 | 20
  No | 99 | 98 | 197
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 22.09 [11.9 to 38.9] | 22.06 [14.5 to 42.2] | 22.08 [11.9 to 42.2]

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Capacity as Measured by 6-minute Walking Distance (6MWD) Month 6 and 12
Description: NOTE: The MAESTRO-OL study was exploratory in nature and no primary efficacy and safety endpoint were defined in the clinical protocol. This and the other exploratory efficacy outcome measures posted were selected to be reported as a primary endpoints. All efficacy analyses were considered exploratory. The analyses of the exploratory efficacy endpoints focused on the absolute values and on the change from DB baseline to Week 16 in the DB study and to Month 6 and Month 12 in the OL study. For missing 6MWD values in the OL study, the following imputation rules were applied: If the reason for missing data was death, a distance of zero (0) meters was imputed for all 6MWD visits from the date of death. For any other reasons, the last available value was carried forward.
Time Frame: From baseline in DB parent study (AC-055-305, NCT01743001) up to month 12 in this OL study.
Measure: Mean (Standard Deviation); unit: meter (m)
Arm/Group | DB-macitentan | DB-placebo
Number analyzed (Participants) | 109 | 108
meter (m)
  6MWD at DB study baseline | 370.6 (74.1) | 381.6 (76.7)
  6MWD at Week 16 in DB study | 395.1 (88.4) | 399.9 (80.6)
  Change in 6MWD from DB study baseline to Week 16 | 24.4 (71.0) | 18.2 (53.0)
  6MWD at Month 6 in OL study | 396.8 (96.5) | 425.0 (72.1)
  Change in 6MWD from DB study baseline to Month 6 | 26.2 (77.9) | 43.4 (51.5)
  6MWD at Month 12 in OL study | 397.1 (103.9) | 421.5 (76.5)
  Change in 6MWD from DB study baseline to Month 12 | 26.5 (79.8) | 39.9 (55.1)

2. Primary Outcome: Change in WHO Functional Class (FC) at Month 6 and 12
Description: Class I: no symptoms with exercise or at rest. No limitation of activity. Class II: No symptoms at rest but slight limitation with ordinary activities causing symptoms (e.g. short of breath with climbing stairs). Class III: may not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. Class IV: symptoms at rest and inability to carry out any physical activity without symptoms. Patients in class IV manifest signs of right heart failure. For missing WHO FC values in the OL study, the following imputation rules were applied: If the reason for missing data was death, class IV was imputed for all WHO visits from the date of death. For any other reasons, the last available value was carried forward.
Time Frame: From baseline in DB parent study (AC-055-305, NCT01743001) up to month 12 in this OL study.
Measure: Count of Participants; unit: Participants
Arm/Group | DB-macitentan | DB-placebo
Number analyzed (Participants) | 109 | 108
Participants
  WHO functional class I at DB study baseline | 0 | 0
  WHO functional class II at DB study baseline | 66 | 65
  WHO functional class III at DB study baseline | 43 | 43
  WHO functional class IV at DB study baseline | 0 | 0
  WHO functional class I at Week 16 in DB study | 3 | 1
  WHO functional class II at Week 16 in DB study | 70 | 77
  WHO functional class III at Week 16 in DB study | 36 | 30
  WHO functional class IV at Week 16 in DB study | 0 | 0
  Improvement from DB study baseline to Week 16 | 10 | 15
  Worsening from DB study baseline to Week 16 | 0 | 1
  WHO functional class I at Month 6 in OL study | 5 | 7
  WHO functional class II at Month 6 in OL study | 74 | 79
  WHO functional class III at Month 6 in OL study | 28 | 22
  WHO functional class IV at Month 6 in OL study | 2 | 0
  Improvement from DB study baseline to Month 6 | 19 | 27
  Worsening from DB study baseline to Month 6 | 3 | 1
  WHO functional class I at Month 12 in OL study | 5 | 7
  WHO functional class II at Month 12 in OL study | 74 | 79
  WHO functional class III at Month 12 in OL study | 28 | 22
  WHO functional class IV at Month 12 in OL study | 2 | 0
  Improvement from DB study baseline to Month 12 | 20 | 31
  Worsening from DB study baseline to Month 12 | 4 | 3

3. Primary Outcome: Change in Borg Dyspnea Score at Month 6 and 12
Description: The Borg dyspnea score rates the severity of dyspnea (difficult or labored breathing) on a scale from 0 ('Nothing at all') to 10 ('Very, very severe - maximal'). For missing Borg dyspnea index values in the OL study, the following imputation rules were applied: If the reason for missing data was death, a value of 10 was imputed for all Borg visits from the date of death. For any other reasons, the last available value was carried forward.
Time Frame: From baseline in DB parent study (AC-055-305, NCT01743001) up to month 12 in this OL study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DB-macitentan | DB-placebo
Number analyzed (Participants) | 109 | 108
score on a scale
  Borg dyspnea score at DB study baseline | 3.0 (1.9) | 2.9 (1.8)
  Borg dyspnea score at Week 16 in DB study | 2.7 (1.9) | 1.9 (1.6)
  Change from DB study baseline to Week 16 | -0.3 (1.4) | -0.2 (1.5)
  Borg dyspnea score at Month 6 in OL study | 2.8 (2.0) | 2.5 (1.8)
  Change from DB study baseline to Month 6 | -0.1 (2.0) | -0.4 (1.5)
  Borg dyspnea score at Month 12 in OL study | 2.9 (2.0) | 2.6 (1.9)
  Change from DB study baseline to Month 12 | -0.1 (2.1) | -0.3 (1.6)

4. Primary Outcome: Change in Peripheral Oxygen Saturation (SpO2) at Rest at Month 6 and 12
Description: No imputation of missing data for SpO2 was applied. Oxygen saturation assessed by pulse oximetry: peripheral oxygen saturation (SpO2) at rest before the 6-minute walk test (6MWT)
Time Frame: From baseline in DB parent study (AC-055-305, NCT01743001) up to month 12 in this OL study.
Population: No imputation of missing data for oxygen saturation as assessed by SpO2 was applied. Therefore out of 109 subjects 104 subjects were analyzed at month 6 and 92 subjects at month 12 in the DB-macitentan group. In the DB-placebo group out of 108 subjects 103 subjects were analyzed at month 6 and 84 subjects at month 12.
Measure: Mean (Standard Deviation); unit: % of oxygen saturation at rest
Arm/Group | DB-macitentan | DB-placebo
Number analyzed (Participants) | 109 | 108
% of oxygen saturation at rest
  SpO2 at DB study baseline | 84.2 (5.6) | 85.4 (5.0)
  SpO2 at Week 16 in DB study | 85.3 (5.8) | 85.6 (5.4)
  Change in SpO2 from DB study baseline to Week 16 | 1.1 (4.0) | 0.2 (4.5)
  SpO2 at Month 6 in OL study: number analyzed (Participants) | 104 | 103
  SpO2 at Month 6 in OL study | 85.9 (5.9) | 87.4 (5.4)
  Change in SpO2 from DB study baseline to Month 6: number analyzed (Participants) | 104 | 103
  Change in SpO2 from DB study baseline to Month 6 | 1.5 (4.9) | 2.0 (4.3)
  SpO2 at Month 12 in OL study: number analyzed (Participants) | 92 | 84
  SpO2 at Month 12 in OL study | 86.4 (6.3) | 87.1 (5.0)
  Change in SpO2 from DB study baseline to Month 12: number analyzed (Participants) | 92 | 84
  Change in SpO2 from DB study baseline to Month 12 | 2.0 (4.4) | 1.6 (4.9)

ADVERSE EVENTS:
Time Frame: From open label study treatment initiation up to 30 days after study treatment discontinuation (max. 24 months + 30 days).
Description: All 217 subjects enrolled in this single-arm open-label (OL) study received 10 mg macitentan to be taken daily and are therefore presented as one group (= all-enrolled analysis set) to report the adverse events in this OL study. From these 217 total subjects 109 received macitentan and 108 placebo in the parent double-blind (DB) study (AC-055-305/MAESTRO, NCT01743001).
Groups:
- All-enrolled Analysis Set: The all-enrolled analysis set includes all subjects enrolled in AC-055-308 / MAESTRO-OL (217 subjects total). All subjects received a film-coated tablet with 10mg mactientan to be taken orally on a daily basis.
Arm/Group | All-enrolled Analysis Set
All-Cause Mortality (participants affected / at risk) | 7/217
Serious Adverse Events (participants affected / at risk) | 62/217
Other Adverse Events (participants affected / at risk) | 152/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-enrolled Analysis Set (N=217)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1)
Antineutrophil cytoplasmic antibody positive (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arterial perforation (Vascular disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Brain abscess (Infections and infestations) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (4)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 2 (2)
Chest pain (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Drug therapy (Surgical and medical procedures) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2)
Retinal artery embolism (Eye disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 6 (7)
Sepsis (Infections and infestations) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-enrolled Analysis Set (N=217)
Bronchitis (Infections and infestations) | 20 (27)
Chest pain (General disorders) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (28)
Diarrhoea (Gastrointestinal disorders) | 18 (20)
Dizziness (Nervous system disorders) | 18 (20)
Fatigue (General disorders) | 11 (11)
Haemoglobin decreased (Investigations) | 20 (29)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 24 (42)
Headache (Nervous system disorders) | 29 (34)
Oedema peripheral (General disorders) | 14 (15)
Upper respiratory tract infection (Infections and infestations) | 61 (119)
Viral upper respiratory tract infection (Infections and infestations) | 21 (35)

LIMITATIONS AND CAVEATS:
The MAESTRO parent study AC-055-305 (NCT01743001) did not meet its primary endpoint. The sponsor decided to prematurely terminate this OL study on January 12th 2018.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related article or abstract written independently by investigators must be submitted to Actelion for review at least 60 days prior to submission for publication or presentation. The list of authors of any formal publication or presentation of study results may include, as appropriate, representatives of Actelion, and will be determined by mutual agreement.

DOCUMENTS (2):
  • Study Protocol (2014-05-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT01739400/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT01739400/SAP_001.pdf